CLINICAL TRIAL: NCT00186069
Title: Randomized, Double Blind Trial of Magnesium Sulfate Tocolysis Versus Intravenous Saline for Suspected Placental Abruption
Brief Title: Magnesium Sulfate vs Placebo for Placental Abruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor of Obstetrics and Gynecology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 79811
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Abruptio Placentae
MeSH Terms: conditions — Abruptio Placentae | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium Sulfate (Active Comparator): Magnesium Sulfate 4 gram bolus, followed by 2 grams per hour
  Interventions: Drug: Magnesium Sulfate
- Normal Saline (Placebo Comparator): Normal Saline 4 gram bolus, followed by 2 grams per hour
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium Sulfate 4 gram bolus, followed by a maintenance dose at 2 grams per hour. Rate increases up to 4 grams per hour may be administered per physician discretion.
  Other Names: Active study drug
  Arms: Magnesium Sulfate
Other: Normal Saline — Normal Saline infusion of 4 gram bolus, followed by 2 grams per hour with rate increases up to 4 grams per hour per physician discretion.
  Other Names: Normal Saline infusion as placebo
  Arms: Normal Saline

SUMMARY:
To evaluate the safety and efficacy of magnesium sulfate for preterm suspected abruption.

DETAILED DESCRIPTION:
We hope to learn if there is a difference in the efficacy of intravenous magnesium sulfate versus intravenous saline infusion in the resolution of vaginal bleeding and contractions in patients with a suspected placental abruption.

ELIGIBILITY:
Inclusion Criteria:

- vaginal bleeding and contractions consistent with suspected placental abruption between 24 and 34 weeks gestation.

Exclusion Criteria:

- preterm labor, severe bleeding necessitating immediate delivery, maternal coagulopathy, fetal distress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2014-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Y El-Sayed, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Colon I, Berletti M, Garabedian MJ, Wilcox N, Williams K, El-Sayed YY, Chueh J. Randomized, Double-Blinded Trial of Magnesium Sulfate Tocolysis versus Intravenous Normal Saline for Preterm Nonsevere Placental Abruption. Am J Perinatol. 2016 Jun;33(7):696-702. doi: 10.1055/s-0036-1571324. Epub 2016 Feb 12. PMID 26871905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium Sulfate | Normal Saline
Started | 15 (Enrollment goal was not reached due to the introduction of magnesium sulfate for neuroprotection) | 15 (Enrollment goal was not reached due to the introduction of magnesium sulfate for neuroprotection)
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate | Normal Saline | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (7.2) | 26.4 (6.3) | 27.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Parity [Number; unit: participants] — Number of women who were nulliparous at enrollment
  participants
    Nulliparous | 2 | 5 | 7
    Multiparous | 13 | 10 | 23
Gestational age at randomization (weeks) [Median (Full Range); unit: weeks of gestation] | 30 [28 to 32] | 30 [25 to 31] | 30 [25 to 32]
Placental location [Number; unit: participants]
  Anterior | 4 | 7 | 11
  Posterior | 9 | 6 | 15
  Fundal | 1 | 2 | 3
  Lateral | 1 | 0 | 1
Vaginal bleeding before study drug administered [Number; unit: participants]
  Mild | 11 | 11 | 22
  Moderate | 4 | 4 | 8
  Heavy | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Undelivered With Resolution of Vaginal Bleeding and Contractions in First 48 Hours
Description: The primary outcome was the proportion of women undelivered at 48 hours with resolution of vaginal bleeding and uterine contractions.
Time Frame: 48 hours after the randomization
Measure: Number; unit: participants
Arm/Group | Magnesium Sulfate | Normal Saline
Number analyzed (Participants) | 15 | 15
participants | 12 | 10
Statistical Analysis 1: Comparison: Magnesium Sulfate vs Normal Saline; Test type: Superiority or Other; p = 0.68, Fisher Exact; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.77 to 1.86]

2. Secondary Outcome: Gestational Age at Delivery (Weeks)
Description: Median gestational age at delivery (in full weeks)
Time Frame: Time of delivery
Measure: Median (Full Range); unit: weeks of gestation
Arm/Group | Magnesium Sulfate | Normal Saline
Number analyzed (Participants) | 15 | 15
weeks of gestation | 36 [32 to 38] | 38 [33 to 39]
Statistical Analysis 1: Comparison: Magnesium Sulfate vs Normal Saline; Test type: Superiority or Other; p = 0.52, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Neonatal Apgar Score at 5 Minutes
Description: The median Apgar score at 5 minutes. Apgar score scale is from 0 to 10 with score 0 expressing the worst neonatal status and score 10 the best status.
Time Frame: At 5 minutes after birth
Measure: Median (Full Range); unit: Apgar score
Arm/Group | Magnesium Sulfate | Normal Saline
Number analyzed (Participants) | 15 | 15
Apgar score | 9 [9 to 9] | 9 [9 to 9]
Statistical Analysis 1: Comparison: Magnesium Sulfate vs Normal Saline; Test type: Superiority or Other; p = 0.95, Fisher Exact

ADVERSE EVENTS:
Time Frame: The adverse events were collected while participants were admitted in labor&delivery and in postpartum units.
Arm/Group | Magnesium Sulfate | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magnesium Sulfate (N=15) | Normal Saline (N=15)
Lethargy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No